CLINICAL TRIAL: NCT02802137
Title: 24-hour Efficacy and Ocular Surface Health With PF Tafluprost and Combined Therapy With PF Tafluprost and Dorzolamide/Timolol Fixed Combination in Open-angle Glaucoma Subjects Insufficiently Controlled With Latanoprost
Brief Title: 24-hour Efficacy and Ocular Surface With Talfuprost and Triple Combined Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor AGP Konstas, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16/5.3.2015
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma; Ocular Surface Disease
Keywords: tafluprost; dorzolamide; timolol; FC
MeSH Terms: conditions — Glaucoma | interventions — tafluprost; dorzolamide; Timolol; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafluprost drops (Active Comparator): Treatment with preservative-free talfuprost drops administered once in the evening. Evaluation of 24-hour efficacy and ocular surface health after 3 months of therapy.
  Interventions: Drug: tafluprost
- Tafluprost and dorzolamide/timolol drops (Active Comparator): Concomitant therapy with preservative-free talfuprost drops administered once in the evening and dorzolamide/timolol fixed combination drops given twice daily. Evaluation of 24-hour efficacy and ocular surface health after 3 months of therapy.
  Interventions: Drug: tafluprost and dorzolamide/timolol

INTERVENTIONS:
Drug: tafluprost
  Other Names: Saflutan, Taflotan
  Arms: Tafluprost drops
Drug: tafluprost and dorzolamide/timolol
  Other Names: Saflutan, Taflotan, Cosopt PF
  Arms: Tafluprost and dorzolamide/timolol drops

SUMMARY:
The study investigated the 24-hour efficacy and ocular surface health with preservative-free tafluprost and a combined preservative-free regimen (tafluprost and dorzolamide/timolol fixed combination) in open-angle glaucoma patients insufficiently controlled on latanoprost monotherapy and showing signs, or symptoms of ocular surface disease with preservative-containing latanoprost monotherapy. This trial randomized open-angle glaucoma patients insufficiently controlled (IOP > 20 mm Hg) on branded, or generic latanoprost monotherapy who required further IOP reduction and who demonstrated clinical signs, or symptoms of ocular surface disease.

ELIGIBILITY:
Inclusion criteria

* Open-angle glaucoma patients (primary open-angle glaucoma, exfoliative, or pigmentary glaucoma) insufficiently controlled on branded, or generic latanoprost monotherapy (IOP > 20 mm Hg as determined by 2 separate IOP measurements at 10:00 ± 1 hour)
* Patients with signs, or symptoms of ocular surface disease.
* Only those open-angle glaucoma subjects who, according to the opinion of the principal investigator, require further IOP reduction.
* Patients must have demonstrated at least 20% IOP reduction at 10:00 (± 1 hour) and who are treated with branded, or generic latanoprost monotherapy for at least 3 months.
* Only subjects with open-angle glaucoma that have exhibited (prior to latanoprost therapy) untreated, sitting IOP evaluated with Goldmann tonometry between 25-39 mm Hg at 10:00 (± 1 hour).
* Age between 21-85 years
* Mild to moderate glaucomatous disc damage and visual field loss (less than -12 dB mean deviation visual field loss attributed to glaucoma
* Those with 0.8 or better vertical cup-to-disc ratio and visual acuity greater than 0.1 in the study eye.
* Open anterior chamber angles.
* Those who have to demonstrate a reliable visual field (at least two visual fields with less than 20% fixation losses, false positives, or negatives)
* Patients who understand study instructions, are willing to attend all follow-up appointments and will comply with study medication usage.

Exclusion criteria

* Patients with a history of less than 10% IOP decrease on any IOP-lowering medication.
* Those with evidence of concurrent conjunctivitis, keratitis, or uveitis in either eye.
* Subjects with a history of inadequate adherence; intolerance, or contraindication to either prostaglandins, β-blockers, dorzolamide, or benzalconium chloride (BAK)
* Patients with severe ocular surface disease, previous intraocular conventional or laser surgery in the study eye (within 6 months prior to enrolment); previous history of ocular trauma; use of corticosteroids (within 3 months before the enrolment) and use of contact lenses.
* Those that on baseline examination show clinical evidence of inflammation, signs of ocular infection (except blepharitis), signs of any corneal abnormality that will affect subsequent IOP measurements
* Subjects that show unwillingness to participate in the trial.
* Females of childbearing potential or lactating mothers.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour efficacy (average intraocular pressure readings over 24 hours) | 3 months

SECONDARY OUTCOMES:
Mean 24-hour peak intraocular pressure | 3 months
Mean 24-hour fluctuation of intraocular pressure | 3 months
Corneal staining | 3 months
Break-up time of tear film | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Chair

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konstas AG, Boboridis KG, Kapis P, Marinopoulos K, Voudouragkaki IC, Panayiotou D, Mikropoulos DG, Pagkalidou E, Haidich AB, Katsanos A, Quaranta L. 24-Hour Efficacy and Ocular Surface Health with Preservative-Free Tafluprost Alone and in Conjunction with Preservative-Free Dorzolamide/Timolol Fixed Combination in Open-Angle Glaucoma Patients Insufficiently Controlled with Preserved Latanoprost Monotherapy. Adv Ther. 2017 Jan;34(1):221-235. doi: 10.1007/s12325-016-0448-9. Epub 2016 Dec 2. PMID 27913991